CLINICAL TRIAL: NCT06598111
Title: Amplifying Consequences to Reduce Dietary Restriction: a Proof-of-Concept Study
Brief Title: Increasing Motivation to Reduce Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Lauren Harris, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00003465
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Restrictive Eating
Keywords: online; experiment; restrictive eating; motivation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Amplified Benefits and Consequences (Experimental): On the first day of the study (day 0), participants in the Amplified Benefits & Consequences condition write a brief, detailed narrative describing a day in their future if they did not restrict their caloric intake and were not concerned about their body weight or shape. Participants type their responses and provide a recording of themselves reading their narrative aloud. On each subsequent day (day 1 through day 6), participants are provided with their written narrative and asked to create a new recording of themselves reading it aloud. After completing their recording and surveys, participants complete a modified version of the Pros and Cons of Anorexia Scale.
  Interventions: Other: Amplified Benefits; Other: Amplified Consequences
- Amplified Benefits (Experimental): On the first day of the study (day 0), participants in the Amplified Benefits condition write a brief, detailed narrative describing a day in their future if they did not restrict their caloric intake and were not concerned about their body weight or shape. Participants type their responses and provide a recording of themselves reading their narrative aloud. On each subsequent day (day 1 through day 6), participants are provided with their written narrative and asked to create a new recording of themselves reading it aloud.
  Interventions: Other: Amplified Benefits
- Amplified Consequences (Experimental): On each day of the study, participants in the Amplified Consequences condition complete the modified Pros and Cons of Anorexia scale and are presented with blurbs about the consequences of restrictive eating.
  Interventions: Other: Amplified Consequences
- Control (Placebo Comparator): Participants in the control condition write a brief narrative considering a future free of concern about finances. As with the active conditions, participants type their narrative on day 0 and record themselves reading it aloud each day.
  Interventions: Other: Control

INTERVENTIONS:
Other: Amplified Benefits — Participants write a brief, detailed narrative describing a day in their future if they did not restrict their caloric intake and were not concerned about their body weight or shape.
  Arms: Amplified Benefits; Amplified Benefits and Consequences
Other: Amplified Consequences — Participants complete the Pros and Cons of Anorexia scale to amplify the consequences of restrictive eating. They are also presented with blurbs about the consequences of restrictive eating.
  Arms: Amplified Benefits and Consequences; Amplified Consequences
Other: Control — Participants write a brief narrative considering a future free of concern about finances.
  Arms: Control

SUMMARY:
The goal of this experiment is to learn how to effectively increase motivation to reduce dietary restriction among young adults engaging in clinically significant restrictive eating. The main questions this study aims to answer are:

* Does imagining a future without restrictive eating increase motivation to reduce restrictive eating?
* Does imagining a future without restrictive eating reduce actual restrictive eating behavior?
* Is it more motivating to think about long-term benefits of reducing dietary restriction, or to focus on short-term consequences of dietary restriction?

Researchers will compare (1) amplifying the possible benefits of reducing restrictive eating, (2) amplifying the negative consequences of restrictive eating, or (3) both is more effective for increasing motivation to reduce dietary restriction over a one-week period.

Participants will:

* Complete daily measures of eating disorder symptoms and motivation for 7 days
* Write a narrative describing a day in the future without restrictive eating and read this narrative aloud daily for 7 days
* Be presented with information regarding the negative consequences of dietary restriction daily for 7 days

DETAILED DESCRIPTION:
This study tests whether amplifying the potential benefits of reducing dietary restriction and/or consequences of maintaining dietary restriction increases motivation to address disordered (i.e., restrictive) eating among college students. This is an online study with a between-groups experimental design which takes place over the course of one week. All study procedures are completed online.

Participants are randomized to one of four conditions: Amplified Benefits & Consequences, Amplified Benefits, Amplified Consequences, or a control condition. Baseline measures are completed on the first day of study enrollment, following randomization to experimental condition. Over the subsequent six days, participants receive daily surveys via email every 24 hours and are given 24 hours to complete each survey. In every condition, participants complete daily self-report measures. Depending on condition, participants also completed the following manipulations:

* Amplified Benefits and Consequences condition: Participants are prompted to write a brief, detailed narrative describing a day in their future if they did not restrict their caloric intake and were not concerned about their body weight or shape. Participants type their responses and provide a recording of themselves reading their narrative aloud. On each subsequent day, participants are provided with their written narrative and asked to create a new recording of themselves reading it aloud. After completing their recording and surveys, participants complete a modified version of the Pros and Cons of Anorexia Scale to amplify the negative consequences of restrictive eating. Next, they read a brief informational blurb about the negative health consequences of restrictive eating.
* Amplified Benefits condition: Participants receive the same narrative prompt and recording instructions as participants in the Amplified Benefits & Consequences condition. They are not asked to complete the modified PCAN or presented with blurbs about the consequences of restrictive eating.
* Amplified Consequences condition: Participants in the Amplified Consequences condition are not prompted to write or record a narrative. After completing daily surveys, they complete the modified PCAN and are presented with blurbs about the consequences of restrictive eating.
* Control condition: Participants write a brief narrative nearly identical Amplified Benefits manipulation; however, their prompt instead asks them to consider a future free of concern about finances. Participants type their narrative and record themselves reading it aloud. Each day, participants create a new recording. Participants in the control condition do not complete the modified PCAN and are not provided with informational blurbs.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Undergraduate student
* Fluent in English
* Engaging in dietary restriction

Exclusion Criteria:

* Engaging in binge eating
* Unable to consent
* Not yet an adult
* Currently pregnant
* Prisoner status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Change in dietary restraint | Baseline (day 0), day 1, day 2, day 3 day 4, day 5, day 6
  Dietary restraint was measured using two items drawn from the Eating Disorder Examination Questionnaire. Each item was rated on a 1-6 scale ranging from 1 (Not at all/never) to 6 (Markedly/all the time). Scores on each item were averaged to create a single dietary restraint score. Changes in daily scores were used to quantify changes in dietary restraint over time.
Change in motivation | Baseline (day 0), day 1, day 2, day 3 day 4, day 5, day 6
  Motivation was measured using the Readiness and Motivation Questionnaire, which is a self-report measure assessing motivation to change disordered attitudes and behaviors. Items reflect four categories: precontemplation, action, internality, and confidence. Respondents rate each item on a percentage scale ranging from zero to 100. The RMQ was modified to include only items assessing dietary restriction, with one item assessing each of the aforementioned categories. Items were anchored to the last 24 hours. Changes in daily scores were used to quantify changes in motivation over time.

SECONDARY OUTCOMES:
Change in body dissatisfaction | Baseline (day 0), day 1, day 2, day 3 day 4, day 5, day 6
  Body dissatisfaction was measured using two items drawn from the Eating Disorder Examination Questionnaire. Each item was rated on a 1-6 scale ranging from 1 (Not at all/never) to 6 (Markedly/all the time). Scores on each item were averaged to create a single body dissatisfaction score. Changes in daily scores were used to quantify changes in body dissatisfaction over time.
Change in shape/weight overvaluation | Baseline (day 0), day 1, day 2, day 3 day 4, day 5, day 6
  Shape/weight overvaluation was measured using three items drawn from the Eating Disorder Examination Questionnaire. Each item was rated on a 1-6 scale ranging from 1 (Not at all/never) to 6 (Markedly/all the time). Scores on each item were averaged to create a single shape/weight overvaluation score. Changes in daily scores were used to quantify changes in shape/weight overvaluation over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Protocol was not designed to allow for IPD sharing.

DOCUMENTS (1):
  • Informed Consent Form (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT06598111/ICF_000.pdf